CLINICAL TRIAL: NCT04193150
Title: Uncontrolled and Possible Severe Asthma in Denmark - What is the Magnitude of the Problem?
Brief Title: Uncontrolled and Possible Severe Asthma in Denmark
Acronym: REASSESS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Kjell Håkansson, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: HVH237-KEJH-REASSESS
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Asthma
Keywords: disease control; socioeconomics; difficult-to-treat
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Induced sputum, Blood samples. Saved in local biobank for future biomarker analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Reassessment Cohort: 150 invited participants in active treatment with high-dose inhaled corticosteroids plus second controller as per NICE guidelines, without active treatment from a pulmonologist.
  Intervention includes:
  1. Extensive pulmonary and allergy assessments. Questionnaires, FeNO-measurement, Skin prick-test, Spirometry, Blood sampling, Body Plethysmography and Diffusion capacity measurement, Bronchial challenge test, Induced sputum.
  2. Treatment optimization As per GINA and Nordic Severe Asthma Network guidelines. Treatment can either be stepped up (e.g. added biological treatment), stepped down or held constant.
  Treatment is then monitored with regard to symptoms and socioeconomical parameteres such as sick leave over a 12 month period using questionnaires and official databases.
  Interventions: Diagnostic Test: Full pulmonary specialist assessment
- Control Cohort: 400 invited participants in active treatment with high-dose inhaled corticosteroids plus second controller as per NICE guidelines, without active treatment from a pulmonologist.
  The control cohort is followed for 12 months using questionnaires and official databases with regard to disease control and socioeconomic parameteres such as sick leave.

INTERVENTIONS:
Diagnostic Test: Full pulmonary specialist assessment — Please see description for the intervention arm.
  Groups: Reassessment Cohort

SUMMARY:
Asthma is a common, chronic disease with a high prevalence in children, adolescents and populations normally fit-to-work. Most asthma patients have a well-controlled disease and thereof a low usage of primary and secondary health care, as well as few sick days. With difficult-to-treat and severe asthma, a much higher health care and sick leave resource usage is seen. Previous studies show that only 1/3rd of patients prescribed high-dose, possibly side effect-laden, medications for difficult-to-treat or possible severe asthma have been seen by a specialist, such as a pulmonologist.

Our study aims to identify socioeconomical patterns and describe patients who are in high dosage asthma treatments, without being seen or treated by a specialist. Furthermore, The Investigators wish to investigate the impact of a systematic pulmonary assessment on quality of life, healthcare utilization and social benefit usage in patients with possible severe asthma.

The results are meant to provide a dataset to identify weaknesses in asthma treatment on a national level, and to lay a foundation for future quality improvements to asthma care in Denmark.

DETAILED DESCRIPTION:
Background & Aim Asthma is the most common chronic disease among children, adolescents and adults. When the diagnosis has been confirmed and the necessary level of treatment established, a well-treated asthma patient is an individual without asthma symptoms. However, asthma is a heterogeneous disease and achieving disease control is far from easy in all asthma patients, although the exact proportion of this problem in real life is unknown. In Denmark, CPR provides the opportunity to track all patients with regard to diagnosis and management, and on a one-by-one basis to merge several informative registers to follow prescribed medication, filled prescriptions, education, area of residence, job, sick leave and referral to secondary care for both asthma and co-morbidities. Based on analysis of data on filled prescriptions from the Danish National Health Service Prescription Database (DNHSPD), it has been demonstrated that only one third of patients classified as having uncontrolled asthma are seen in secondary care.

Based on a nationwide asthma database and clinical confirmation, The Investigators aim to:

* Describe the patient demographics and disease-burden in patients with possible hidden severe asthma in Denmark, using the national databases.
* Elucidate the real-world prevalence of hidden severe asthma in Denmark, by systematic assessment of patients with possible hidden severe asthma.
* Investigate the impact of systematic asthma assessment on quality of life and asthma control in patients with possible hidden severe asthma.

Hypotheses & Expected results

1. Within the last year, a large proportion of asthma patients (75%) prescribed medium to high doses of inhaled corticosteroids (ICS) have not had their lung function measured, had no new asthma drugs prescribed and have not been referred to secondary care for further assessments.
2. A significant number of asthma patients in primary care are prescribed high doses of ICS and filled prescriptions for >200 puffs of rescue medication (short-acting beta 2-agonists (SABA) or anticholinergics (SAMA)) per year over a period of 2 years, exhibiting low disease awareness of the difficult to manage asthma patients by both doctors and patients.
3. In primary care, more than 75% of asthma patients prescribed high dose ICS and a second controller have been seen in secondary care within the last year, leaving few (25%) with possible hidden severe asthma in primary care.
4. In primary care, there is a significant mismatch between general practitioner (GP)-based diagnosis of severe asthma (based on prescription data) and the true prevalence of severe asthma following guideline-based systematic assessment for severe asthma.
5. A systematic pulmonary assessment in patients with possible severe asthma leaves few with a severe asthma diagnosis and increases disease control in patients with moderate-to-mild asthma. A significant proportion of patients are able to step-down in inhaled steroid treatment as described in GINA guidelines.

Methods

The initial studies are designed as retrospective, observational studies with a real-world evidence, registrybased design. The study period is 1/6-14 to 31/5-18. Databases used are:

* Danish Clinical Registries (DCR) - Asthma
* National Patient Registry (NPR) & Statistics Denmark (DST)
* The Danish National Health Service Prescription Database (DNHSPD)

The clinical follow-up (reassessment) study is designed as an interventional, non-randomized, non-blinded clinical study with the aim of assessing the effect of systematic asthma assessment (as suggested by the Nordic Severe Asthma Network) on patients with possible severe asthma not seen by a pulmonologist.

Effects are measured as

1. improvements of symptoms and quality of life according to questionnaires and
2. improvements of clinical variables such as lower peak expiratory flow (PEF) variability.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-74 at the time of signing the informed consent form.
2. Physician diagnosed asthma.
3. Active treatment

   1. Defined as minimum 1 filled prescription of an obstructive pulmonary disease drug (ACT R03) during the last 12 months.
   2. Dosage of ICS as described in the NICE guidelines.
4. No asthma-related contact to a respiratory medicine outpatient clinic during the last 36 months.

Exclusion Criteria:

1. Inability to give informed consent.
2. Inability to participate in questionnaires during the 12 months follow-up. Note: follow-up questionnaires can be provided in printed form, should the patient not have internet access.
3. Inability to participate in baseline spirometry, blood sampling and skin prick test.
4. Inability to abstain from pre-assessment meals and caffeine (2 hours), smoking (same day), ICS (1 day) and bronchodilators (24 hours).
5. Any clinically important concomitant severe pulmonary disease such as COPD without an asthmatic/significant reversible component, pulmonary fibrosis, cystic fibrosis, lung cancer, previous lobectomy, alpha 1 anti-trypsin deficiency, primary ciliary dyskinesia, allergic aspergillosis, eosinophilic granulomatosis with polyangiitis, hypereosinophilic syndrome.

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruitment to the reassessment study is performed through the national Danish Clinical Registries - Asthma-database, which consists of about 200 000 patients. Patients in the database have either 1) had specialist treatment for their asthma or 2) redeemed prescriptions for asthma medications such as inhaled corticosteroids.
  The population sought is a representative sample of patients who are receiving high-dosage inhaled corticosteroid treatment for their asthma by their general practitioner.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of severe asthma | 12 months
  The actual prevalence of severe asthma in a cohort of asthma patients treated with high-dose inhalation corticosteroids by a general practitioner.

SECONDARY OUTCOMES:
Asthma Control Test/Astma Control Questionnaire-scores | 12 months
  Changes in Asthma Control Test/Astma Control Questionnaire-scores over time and after pulmonary specialist reassessment
  Asthma Control Test is a 5 question questionnaire on asthma disease symptom burden, ranging from 5 to 25, with scores under 20 being indicative of poor disease control, and scores between 20 and 25 indicating some or full disease control.
  Astma Control Questionnaire is a 7 item questionnaire on asthma diease symptom burden, rescue medication use and lung function. Each item is scored from 0 to 6, with a mean score (total score of all items divided by 7) of 0 to 0.75 suggesting well controlled disease, 0.76-1.5 is a "gray area" and >1.5 is indicative of poorly controlled disease.
SABA/SAMA usage | 12 months
  Change in redemption of short-acting bronchodilator prescriptions as a surrogate for increased disease control
Exposure to systemic corticosteroids | 12 months
  Change in redemption of systemic corticosteroid prescriptions as a surrogate for increased disease control.
Acute exacerbations | 12 months.
  Change in number of exacerbations requiring systemic corticosteroids or hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suppli Ulrik, Professor, Study Chair — csulrik@dadlnet.dk

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing upon reasonable request, however, approval from Statistics Denmark and the National Prescription Database might be required.